CLINICAL TRIAL: NCT02972359
Title: Open-label Safety Trial of Intravenous Neridronic Acid in Subjects With Complex Regional Pain Syndrome (CRPS)
Brief Title: Safety of Intravenous Neridronic Acid in CRPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF7013-03; 2016-001164-11 (EudraCT Number); U1111-1180-8099 (Other: World Health Organization)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Neridronic Acid; Neridronate; CRPS; RSD (reflex sympathetic dystrophy)
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neridronic acid (Experimental): Neridronic acid 100 mg administered on Day 1, Day 4, Day 7, and Day 10, resulting in a total dose of neridronic acid 400 mg.
  Interventions: Drug: Neridronic acid

INTERVENTIONS:
Drug: Neridronic acid — Neridronic acid administered as intravenous infusion.

SUMMARY:
The aim of this trial was to investigate the safety of intravenous neridronic acid in patients with complex regional pain syndrome (CRPS).

The trial was divided into 3 periods: a 60-day enrollment period, a treatment period consisting of 4 infusions over 10 days, and a follow-up period of approximately 50 weeks (with visits at Week 2, Week 6, Week 12, Week 26, Week 39, and Week 52).

DETAILED DESCRIPTION:
At the Enrollment Visit the trial objectives, procedures, and risks were explained to the participants and the informed consent form was signed. Medical history was obtained, a physical examination was conducted, and other safety assessments were performed. Signs and symptoms of CRPS were assessed to confirm the diagnosis of CRPS according to the Budapest clinical criteria. Participants were trained to report their pain. Calcium and vitamin D supplementation were initiated to ensure sufficient vitamin D levels prior to treatment.

Participants meeting all eligibility criteria received infusions of investigational medicinal product (IMP) during visits on Day 1, Day 4, Day 7, and Day 10. Flexibility of ±1 day was allowed for Day 4, Day 7, and Day 10 whilst ensuring a minimum period of 48 hours between infusions. During the treatment period and follow-up period, pain intensity ratings were captured at the site visits in a patient reported-outcome system.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Male or female participant at least 18 years of age at Visit 1.
* A diagnosis of complex regional pain syndrome according to the clinical diagnostic criteria recommended by the International Association for the Study of Pain (IASP; "Budapest clinical criteria"), assessed at Visit 1. Signs and symptoms of CRPS must apply to an affected limb (arm or leg) and must demonstrate asymmetry with respect to the contralateral limb.
* Ongoing moderate to severe chronic pain, including a baseline current pain intensity score of greater than or equal to 4 using an 11-point Numerical Rating Scale, referring to the CRPS-affected limb, at Visit 2 (prior to dosing).
* In stable treatment and follow-up therapy for CRPS for at least 1 month prior to allocation to treatment (Visit 2). Participants must have failed trials of at least 2 treatments for CRPS, one of which must be a pharmacologic treatment.
* Women of child-bearing potential must have a negative urine beta-human chorionic gonadotropin (β-HCG) pregnancy test at Visit 1 and must be using 2 forms of medically acceptable contraception, including at least 1 highly effective method of contraception with a low failure rate, defined as less than 1% per year (e.g., oral contraceptives or intrauterine device), and a second medically acceptable method such as use of condoms with spermicide by their male partner. A barrier method alone is not acceptable. Highly effective methods of contraception must be used for at least 1 month prior to Visit 2 and for the duration of the trial.
* Participants must be able to communicate meaningfully, be able to differentiate with regard to location and intensity of the pain, and be able to answer the questions in the questionnaires used in this trial (assistance in filling out the questionnaires may be provided, if required due to motor or other impairment).

Exclusion Criteria:

* Evidence of renal impairment (estimated glomerular filtration rate [eGFR] less than 60 mL/min/1.73 m2 using the 2009 Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] creatinine equation [Levey et al. 2009] or a urinary albumin creatinine ratio greater than 150 mg/g), based on central safety laboratory data obtained prior to Visit 2, or a history of chronic kidney disease. Note: a single repeat laboratory test is allowed.
* Serum calcium or magnesium outside of the central laboratory's reference range, based on central safety laboratory data obtained prior to Visit 2 (a single repeat laboratory test is allowed); a history of hypocalcemia or a metabolic disorder anticipated to increase risk for hypocalcemia (e.g., hypoparathyroidism); concomitant use of drug(s) with known potential to cause hypocalcemia (e.g., aminoglycosides).
* Vitamin D deficiency, defined as a 25(OH)D level less than 30 ng/mL, based on central safety laboratory data obtained prior to Visit 2 (up to 4 repeat laboratory tests are allowed). Participants with vitamin D deficiency should receive appropriate supplementation during the enrollment period. A vitamin D level of at least 30 ng/mL must be documented prior to allocation to investigational medicinal product (IMP).
* Corrected QT interval (according to Fridericia's formula; QTcF) greater than 470 ms (average of 3 electrocardiograms [ECGs] obtained at Visit 1); serum potassium outside the central laboratory's reference range at Visit 1; clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or an indwelling pacemaker; evidence of complete left bundle branch block; complete atrioventricular block; history of Long QT Syndrome or a relative with this condition; or any other known risk factor for torsade de pointes.
* Participants receiving medications with a known risk of torsades de pointes within 7 days prior to allocation. Participants receiving selective serotonin re-uptake inhibitor antidepressants (e.g., citalopram, escitalopram) or tricyclic antidepressants are eligible if the QT-interval values do not meet the exclusion criteria, the medication was started at least 1 month prior to allocation, the dose is stable, and the dose is anticipated to remain stable until at least 4 days after the last infusion of IMP.
* Anticipated requirement for treatment with oral or intravenous bisphosphonate for another condition such as osteoporosis during the trial, or administration of denosumab (Prolia®) or other drugs affecting bone turnover or bone metabolism within 6 months prior to Visit 1.
* History of any allergic or hypersensitivity reaction to neridronic acid or other bisphosphonate, acetaminophen, or to vitamin D or calcium supplements.
* Recent tooth extraction or other invasive dental procedure (within 3 months prior to Visit 1), unhealed or infected extraction site, or significant dental/periodontal disease (e.g., impacted molars, severe tooth decay, foci of infection) that may predispose to need for tooth extraction or other invasive dental procedures during the trial. Participants with indeterminate, suspicious or unreliable dental history, in the opinion of the investigator, must undergo a dental examination prior to receiving treatment.
* Evidence of denture-related gum trauma or improperly fitting dentures causing injury.
* Prior radiation therapy of the head or neck (within 1 year of Visit 1).
* History of malignancy within 2 years prior to Visit 1, with the exception of basal cell carcinoma.
* Use of nerve blocks, ketamine infusions, intravenous immunoglobulin, acupuncture, electromagnetic field treatment, or initiation/implementation of radiofrequency ablation or other sympathectomy procedures, or peripheral nerve stimulation within 6 weeks prior to Visit 2.
* Evidence of current alcohol or drug abuse, or history of alcohol or drug abuse within 2 years of Visit 1, based on participant history and physical examination and according to the investigator's judgment.
* Any other severe medical condition, including severe depression, or any other severe mood disorder, that in the opinion of the investigator may affect efficacy or safety assessments or may compromise the participant's safety during trial participation.
* Women who are pregnant or breastfeeding.
* Elevated aspartate aminotransferase or alanine aminotransferase greater than 2-fold upper limit of normal, based on central safety laboratory data obtained at Visit 1, or current evidence of chronic liver disease. Safety laboratory testing may be repeated prior to Visit 2, and participants will be allowed in the trial if results of 2 consecutive tests, at least 3 days apart, are less than or equal to 2-fold upper limit of normal.
* Participation in another investigational drug trial within 3 months prior to Visit 1 or any previous trial with neridronic acid, with the exception of participants of KF7013-01 who were assigned to placebo and did not receive neridronic acid.
* Participant is engaged in litigation related to their disability from CRPS in which monetary gain or loss (or other compensation) may affect their objective participation in the trial.
* Participants taking forbidden concomitant medications/therapies or not being able to follow the rules of use of concomitant treatment.
* Participants incapable of signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (46):
- United States (42):
  - US017: Cactus Clinical Research, Inc., Phoenix, Arizona
  - US028: Quality of Life Medical and Research Centers LLC, Tucson, Arizona
  - US045: Woodland International Research Group, Little Rock, Arkansas
  - US044: Woodland Research Northwest, Rogers, Arkansas
  - US012: Orange County Research Institute, Anaheim, California
  - US022: Core Healthcare Group, Cerritos, California
  - US033: Alliance Research Centers, Laguna Hills, California
  - US027: The Helm Center for Pain Management, Laguna Woods, California
  - US003: Samaritan Center for Medical Research, Los Gatos, California
  - US010: Catalina Research Institute, LLC, Montclair, California
  - US014: Northern California Research, Sacramento, California
  - US034: Mountain View Clinical Research, Inc., Denver, Colorado
  - US032: South Lake Pain Institute, Clermont, Florida
  - US001: Sunrise Research Institute, Inc, Miami, Florida
  - US046: AMPM Research Clinic, Miami, Florida
  - US035: Compass Research, Orlando, Florida
  - US031: Gold Coast Research, LLC, Plantation, Florida
  - US011: Clinical Research of West Florida, Inc., Tampa, Florida
  - US040: Palm Beach Research Center, West Palm Beach, Florida
  - US026: Better Health Clinical Research Inc., Newnan, Georgia
  - US004: Northwestern University - Feinberg School of Medicine - Rehabilitation Institute of Chicago (RIC), Chicago, Illinois
  - US036: University Anesthesiologists, S.C., Chicago, Illinois
  - US029: Great Lakes Clinical Trials LLC, Chicago, Illinois
  - US005: International Clinical Research Institute, Overland Park, Kansas
  - US037: St. Louis Clinical Trials, LC, St Louis, Missouri
  - US051: Creighton University, Osteoporosis Research Center, Omaha, Nebraska
  - US002: Princeton Medical Institute, Princeton, New Jersey
  - US049: Premier Pain Centers, LLC, Shrewsbury, New Jersey
  - US048: Albany Medical College, Albany, New York
  - US043: Translational Pain Research, University of Rochester, Rochester, New York
  - US009: The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - US016: North Star Medical Research, LLC, Middleburg Heights, Ohio
  - US007: Medical Research International, Oklahoma City, Oklahoma
  - US006: Abington Neurological Associates, LTD., Willow Grove, Pennsylvania
  - US020: Clinical Trials of South Carolina, Charleston, South Carolina
  - US038: Vanderbilt University Medical Center, Nashville, Tennessee
  - US019: Austin Center for Clinical Research, Austin, Texas
  - US008: Pioneer Research Solutions, Houston, Texas
  - US023: Axios Research, LLC, Salt Lake City, Utah
  - US018: Washington Center for Pain Management, Bellevue, Washington
  - US015: Northwest Clinical Research Center, Bellevue, Washington
  - US013: Swedish Pain Services/ Research Institute, Seattle, Washington
- Germany (4):
  - DE001: Klinische Forschung Hannover-Mitte GmbH, Hanover
  - DE004: Schmerzambulanz Medizinishe Hochschule Hannover, Hanover
  - DE006: AmBeNet GmbH, Leipzig
  - DE002: Schmerztagesklinik der Anästhesiologie Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 20 December 2016.
Pre-assignment Details: A total of 580 participants signed an informed consent form, 318 participants hereof were allocated to treatment. Two of the allocated participants did not meet inclusion criteria/met exclusion criteria, thus 316 participants received treatment.
Groups:
- Neridronic Acid: Neridronic acid 100 mg administered on Day 1, Day 4, Day 7, and Day 10, resulting in a total dose of neridronic acid 400 mg as intravenous infusion.
Period: Overall Study
Arm/Group | Neridronic Acid
Started | 318
Completed | 247
Not Completed | 71
Not completed — Incl. criteria not met/Exclusion met | 2
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 30
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 26
Not completed — Other reasons | 5
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 290
  >=65 years | 26
Age, Continuous [Mean (Full Range); unit: years] | 47.4 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 300
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 297
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 308
  Germany | 8
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (7.4)
Baseline current pain intensity 11-point NRS [Mean (Standard Deviation); unit: units on a scale] — Measured using an 11-point Numerical rating scale (NRS) by answering the following question: "Please rate your pain by selecting the one number that best describes how much pain you have right now." Scores ranged from 0 (no pain) to 10 (pain as bad as you can imagine), a higher score indicates more pain. Baseline was the score assessed before the first dose of investigational medicinal product (IMP). Population: One participant's baseline pain assessment was missing (N=315). Full Analysis Set
  units on a scale
    number analyzed (Participants) | 315
    (all) | 6.59 (1.58)
Baseline Pain Interference score of the Brief Pain Inventory (BPI) [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Brief Pain Inventory (BPI) Interference Scale questionnaire, which measures the impact of pain on functioning and well-being. The 7 pain interference items: general activity, walking, work, mood, enjoyment of life, relations with others, and sleep, are each rated on a 0 to 10 scale using a 24-hour recall period, with 0 indicating "does not interfere" and 10 indicating "completely interferes". The total Pain Interference Score is calculated by adding the scores for the 7 questions and dividing by 7. This gives an interference score with a range from 0 to 10. Population: 20 participants baseline pain assessment were missing. Full Analysis Set
  units on a scale
    number analyzed (Participants) | 296
    (all) | 7.3 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Occurrence of Any Treatment Emergent Adverse Event (TEAE)
Description: The primary endpoint of this trial was a binary endpoint assessing whether or not a participant experienced any TEAE.
Time Frame: Day 1 to Week 52
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
Participants
  Participants with TEAE | 277
  Participants with serious TEAE | 27
  Participants with non-serious TEAE | 275
  Participants with unexpected TEAE | 267
  Participants with related TEAE | 190
  Participants with related serious TEAE | 3
  Participants with TEAE leading to IMP discont. | 12
  Participants with TEAE leading to trial discont. | 6

2. Secondary Outcome: Number of Participants With Occurrence of Permanent Discontinuation From Treatment Due to an Adverse Event
Description: The investigator could choose to permanently discontinue a participant from treatment if continued exposure of the participant to neridronic acid could have posed an undue risk to the participant.
Time Frame: Day 1 to Day 10
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
Participants | 12

3. Secondary Outcome: Change From Baseline in the Current Pain Intensity Score
Description: The current Complex Regional Pain Syndrome (CRPS)-related pain intensity score was captured at each visit using an 11-point numerical rating scale where 0 = "no pain" and 10 = "pain as bad as you can imagine", a higher score indicates more pain.
Time Frame: Baseline to Week 12 and Week 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
units on a scale
  Baseline to Week 12: number analyzed (Participants) | 283
  Baseline to Week 12 | -1.54 (2.27)
  Baseline to Week 26: number analyzed (Participants) | 269
  Baseline to Week 26 | -1.57 (2.45)

4. Secondary Outcome: Number of Participants With Response to Treatment, Defined as at Least 30% Decrease From Baseline in the Current Pain Intensity Score
Description: Participants with at least a 30 percent decrease in the current pain intensity score were considered to have responded to treatment.
Time Frame: Baseline, at Week 12 and Week 26
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
Participants
  At least 30% pain reduction - Week 12 | 105
  At least 30% pain reduction - Week 26 | 110

5. Secondary Outcome: Number of Participants With Response to Treatment, Defined as at Least 50% Decrease From Baseline in the Current Pain Intensity Score
Description: Participants with at least a 50 percent decrease in the current pain intensity score were considered to have responded to treatment.
Time Frame: Baseline, at Week 12 and Week 26
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
Participants
  At least 50% pain reduction - Week 12 | 75
  At least 50% pain reduction - Week 26 | 74

6. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12
Description: The Patient Global Impression of Change (PGIC) is a self-reported measure of perceived change in overall condition since the start of the study. Participants selected one of seven responses ranging from "very much improved" to "very much worse". A response of "very much improved" or "much improved" is generally regarded as a clinically important improvement.
Time Frame: at Week 12
Population: Full Analysis Set; 286 out of 316 participants attended the visit at Week 12 and were asked to complete the PGIC questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 286
Participants
  Very Much Improved | 31
  Much Improved | 71
  Minimally Improved | 98
  No Change | 45
  Minimally Worse | 23
  Much Worse | 12
  Very Much Worse | 3
  Missing | 3

7. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 26
Description: as for outcome 6
Time Frame: at Week 26
Population: Full Analysis Set; 273 out of 316 participants attended the visit at Week 26 and were asked to complete the PGIC questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 273
Participants
  Very Much Improved | 38
  Much Improved | 58
  Minimally Improved | 84
  No Change | 52
  Minimally Worse | 25
  Much Worse | 10
  Very Much Worse | 2
  Missing | 4

8. Secondary Outcome: Change in the Pain Interference Score of the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) Interference Score is the mean value of 7 self-reported items in question 9 of the BPI Short Form Questionnaire. Participants rated their interference of pain with general activity, walking, work, sleep and other activities in the past 24 hours, with possible ratings from 0 (does not interfere) to 10 (completely interferes). The BPI interference Score ranges from 0 to 10, with higher values indicating greater pain interference of daily activities.
Time Frame: Baseline to Week 12 and Week 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neridronic Acid
Number analyzed (Participants) | 316
score on a scale
  Baseline to Week 12: number analyzed (Participants) | 264
  Baseline to Week 12 | -2.2 (2.49)
  Baseline to Week 26: number analyzed (Participants) | 251
  Baseline to Week 26 | -2.1 (2.64)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 52
Description: 318 participants were allocated to treatment. Two participants did not meet inclusion criteria/met exclusion criteria, thus 316 participants were treated (Safety Set).
  Participants were questioned about possible adverse events with non-leading questions before administration of the IMP and at regular intervals thereafter. All adverse events reported spontaneously by participants at any time point were also documented.
  Treatment emergent adverse events are reported.
Arm/Group | Neridronic Acid
All-Cause Mortality (participants affected / at risk) | 1/316
Serious Adverse Events (participants affected / at risk) | 27/316
Other Adverse Events (participants affected / at risk) | 275/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neridronic Acid (N=316)
Angina unstable (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Condition aggravated (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neridronic Acid (N=316)
Headache (Nervous system disorders) | 65 (96)
Myalgia (Musculoskeletal and connective tissue disorders) | 52 (70)
Nausea (Gastrointestinal disorders) | 34 (46)
Fatigue (General disorders) | 32 (39)
Condition aggravated (General disorders) | 30 (44)
Pain (General disorders) | 28 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (30)
Pyrexia (General disorders) | 18 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 17 (20)

LIMITATIONS AND CAVEATS:
Due to the open-label, uncontrolled nature of the trial and the concomitant use of pain medication, the effect of neridronic acid on pain intensity and the side effect profile of neridronic acid have to be interpreted with care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party (e.g., the sponsor, the coordinating investigator) has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02972359/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02972359/SAP_001.pdf